CLINICAL TRIAL: NCT00341913
Title: Network on Antimicrobial Resistance in Staphylococcus Aureus
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999900012; OH00-I-N012
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-17

CONDITIONS: Staphylococcus Aureus
Keywords: Research; Repository; Registry; Surveillance; Databases
MeSH Terms: conditions — Staphylococcal Infections

SUMMARY:
Reduced susceptibility of Staphyloccus aureus to the glycopeptide antibiotic vancomycin is causing increasing concern worldwide in view of the threat of increased morbidity and mortality caused by such resistant organisms. MRL Pharmaceutical Services, a Division of Focus/MRL, has been contracted by NIAID to establish a Network on Antimicrobial Resistance in S. aureus (NARSA) to document cases where staphylococcal isolates with reduced susceptibility to vancomycin (MIC's greater than or equal to 4 micrograms/ml) have arisen and to procure such isolates into a central repository for distribution to registered approved researchers.

MRL will be responsible for contacting sites where such isolates have been reported to discuss the test methods used to determine the reduced vancomycin susceptibility status of the isolate. Once the MRL Laboratory has determined that the isolate meets the criteria stated above, the site will be asked to ship the isolate to MRL as a possible candidate for inclusion in the NARSA Repository. The procurement strategy will involve issuing each isolate a temporary strain designation number which will be destroyed once the antibiotic profile of the isolate has been confirmed at MRL, thus preventing any link to the data generated by the site. The isolate and its antimicrobial susceptibility profile to several key drugs will be recorded in the NARSA Repository database. Demographic information related to the isolate and collected from the site includes: The Name of the Donor Site/Institution, City (to be held in a separate secured database, these data points are not available to registered user); State, Country of Donor Site; Isolation Date; Age; Sex; Patient Location; Patient Service; Culture Source; Reporting History. This information will be held in the Registry database. Since patient-specific information will not be collected, a request for a waiver of informed consent has been requested herein.

NIAID funded investigators (NARSA Core Investigators) and other approved registered users whose research focuses on S. aureus will have access to the Registry/Repository database and will be able to request isolates for use in their research. Facility specific information will be held in a separate secured database that is not available to registered researchers unless approved through an IRB review.

DETAILED DESCRIPTION:
Reduced susceptibility of Staphyloccus aureus to the glycopeptide antibiotic vancomycin is causing increasing concern worldwide in view of the threat of increased morbidity and mortality caused by such resistant organisms. MRL Pharmaceutical Services, a Division of Focus/MRL, has been contracted by NIAID to establish a Network on Antimicrobial Resistance in S. aureus (NARSA) to document cases where staphylococcal isolates with reduced susceptibility to vancomycin (MIC's greater than or equal to 4 micrograms/ml) have arisen and to procure such isolates into a central repository for distribution to registered approved researchers.

MRL will be responsible for contacting sites where such isolates have been reported to discuss the test methods used to determine the reduced vancomycin susceptibility status of the isolate. Once the MRL Laboratory has determined that the isolate meets the criteria stated above, the site will be asked to ship the isolate to MRL as a possible candidate for inclusion in the NARSA Repository. The procurement strategy will involve issuing each isolate a temporary strain designation number which will be destroyed once the antibiotic profile of the isolate has been confirmed at MRL, thus preventing any link to the data generated by the site. The isolate and its antimicrobial susceptibility profile to several key drugs will be recorded in the NARSA Repository database. Demographic information related to the isolate and collected from the site includes: The Name of the Donor Site/Institution, City (to be held in a separate secured database, these data points are not available to registered user); State, Country of Donor Site; Isolation Date; Age; Sex; Patient Location; Patient Service; Culture Source; Reporting History. This information will be held in the Registry database. Since patient-specific information will not be collected, a request for a waiver of informed consent has been requested herein.

NIAID funded investigators (NARSA Core Investigators) and other approved registered users whose research focuses on S. aureus will have access to the Registry/Repository database and will be able to request isolates for use in their research. Facility specific information will be held in a separate secured database that is not available to registered researchers unless approved through an IRB review.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

This study is concerned with the collection of data on the antimicrobial phenotypes of bacterial isolates and not the patient(s) from which they were isolated. Therefore, criteria for the inclusion or exclusion of patients does not apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-03-16; Study Completion 2008-06-17

CONTACTS AND LOCATIONS:
Locations (1):
- MRL Pharmaceutical Services, Herndon, Virginia, United States